CLINICAL TRIAL: NCT03878537
Title: Recurrence Monitoring in NSCLC Using Circulating Tumor DNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Scripps Health (Other); Lexent Bio, Inc. (Industry)
Responsible Party: Principal Investigator, Aditya Sarvaria, MD, Investigator, Scripps Translational Science Institute
Other Study IDs: IRB-17-7057
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research study is investigating the role of cell free tumor DNA profiling in determining disease relapse and/or progression for patients with advanced NSCLC.

DETAILED DESCRIPTION:
The objective of this study is to determine the ability of cell free tumor DNA genomic profiling to predict disease relapse or progression while on therapy for advanced stage NSCLC in comparison to current standard objective measures of disease relapse or progression.

This study is a prospective observational study. The investigators will assess whole genome sequencing from patient blood samples collected alongside routine blood draws with each treatment cycle to determine the tumor load score at each timepoint while on therapy. CT images will be obtained at routinely ordered timepoints throughout therapy and will be used in the assessment for standard clinical or radiographic evidence of disease progression. These methods of measuring disease progression will be compared in a lead time analysis.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve biopsy confirmed not surgically resectable stage III or greater NSCLC
* Baseline CT imaging available

Exclusion Criteria:

* Patients unable to undergo biopsy for initial tissue diagnosis
* Patients who do not wish to pursue standard of care therapy
* Patients with another diagnosis of malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 or older with NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-03-14 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 24 months
  Cell free tumor DNA based PFS
Progression Free Survival | 24 months
  Clinical or radiographic based PFS

CONTACTS AND LOCATIONS:
Overall Officials: Marin Xavier, Principal Investigator — Scripps Health
Locations (1):
- Scripps Health/Scripps Clinic Hillcrest/Scripps Clinic Torrey Pines, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No